CLINICAL TRIAL: NCT03778476
Title: Isometric Exercise and Endogenous Pain Modulation
Brief Title: Isometric Exercise and Endogenous Pain Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HR3035
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Fibromyalgia
Keywords: Exercise; pain sensitivity; fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The two groups will participate in two sessions receiving intervention or no intervention in a randomized manner.
Who Masked: Participant
Masking Description: The participant is masked to the hypotheses of the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isometric Exercise (Experimental): Participants will perform a submaximal voluntary contraction of the quadriceps muscle to task failure.
  Interventions: Other: Isometric Exercise
- Quiet Rest (No Intervention): Participants will sit quietly for a period of time that mimics the exercise.

INTERVENTIONS:
Other: Isometric Exercise — Participants will be asked to hold a submaximal voluntary contraction of the quadriceps muscle as long as they can (task failure).
  Arms: Isometric Exercise

SUMMARY:
The purpose of this study is to identify the acute effects of isometric exercise on the inhibition of pain in individuals with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a chronic pain condition that is characterized by widespread pain which affects 5-8% of the general population. Past research has shown that people with FMS demonstrate enhanced pain facilitation and reduced pain inhibition in the central nervous system. Incorporating a biopsychosocial model of pain may help develop strategies to prevent the functional decline and alleviate the suffering that occurs in this population. Exercise is a mainstay of pain rehabilitation with multiple health benefits, one of which is decreasing pain; a phenomenon known as exercise induced hypoalgesia (EIH). Emerging evidence has shown that exercise decreases pain facilitation in healthy adults and in some individuals with FMS. However, it's unclear whether exercise improves pain inhibition in individuals with FMS. The purpose of this study is to investigate endogenous pain inhibition, measured by conditioned pain modulation (CPM), following isometric exercise of the quadriceps muscle in individuals with FMS. In addition, factors that might affect this response such as physical activity, body composition, and psychosocial issues will be examined. Understanding how exercise impacts pain and the contributing factors will help guide the prescription of exercise to optimize pain rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-75 diagnosed with fibromyalgia or healthy controls will be included in the study.

Exclusion Criteria:

* cardiovascular disease, cancer, pregnancy, arthritis, diabetes, claustrophobia, Reynaud's disease, osteoporosis, neuropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Conditioned Pain Modulation | baseline, immediately after exercise or quiet rest
  the change in pressure pain threshold (kPa) during or after the immersion of the foot in a cold water bath (approximately 6 degrees) compared with baseline (before foot submersion) constitutes the measure of conditioned pain modulation in this study.

SECONDARY OUTCOMES:
Vibration Perception Threshold | baseline, immediately after exercise or quiet rest
  a biothesiometer will be used to measure sense of vibration (threshold) local and distal from the exercising muscle.

OTHER OUTCOMES:
Numerical Pain Rating Scale (NPRS) | baseline, during exercise, and immediately after exercise or quiet rest
  in both sessions, pain intensity will be evaluated during ice water bath immersion (i.e. before and after exercise or quiet rest) and during exercise using an 11-point NPRS with 0 being no pain and 10 worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Hoeger Bement, PT, PhD, Principal Investigator — Marquette University; Ali Alsouhibani, PT, MS, Study Director — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States